CLINICAL TRIAL: NCT06641362
Title: Pivotal Clinical Study of VDI's Ultra-High Frequency Electrocardiogram (UHF-ECG) for the Diagnosis of Ventricular Electrical Dyssynchrony (VED): THE SYNC Study
Brief Title: Ultra-High Frequency - Electrocardiogram (UHF-ECG) for the Diagnosis of Ventricular Electrical Dyssynchrony (VED)
Acronym: SYNC
Status: Recruiting | Type: Observational
Sponsor: VDI Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN001
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Bradycardia; Heart Failure; Ventricular Dysfunction
MeSH Terms: conditions — Bradycardia; Heart Failure; Ventricular Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment Group: Participant controlled with standard ECG measurement and VDI UHF-ECG measurement both taken sequentially.
  Interventions: Device: Ultra High Frequency Electrocardiogram (UHF-ECG)

INTERVENTIONS:
Device: Ultra High Frequency Electrocardiogram (UHF-ECG) — Electrocardiograms used on participants scheduled to undergo pacemaker implantation for bradycardia and/or heart failure.
  Other Names: Standard 12 lead Electrocardiogram (ECG)

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of the VDI UHF-ECG System in the diagnosis of ventricular dyssynchrony when compared to the 12-lead ECG in patients with bradycardia and heart failure indicated for pacemaker implantation.

ELIGIBILITY:
Inclusion Criteria:

* Adults with bradycardia scheduled for pacemaker implant or heart failure patients indicated for cardiac resynchronization therapy (CRT) with one of the following:

  * Bradycardia with ventricular synchrony and QRS duration < 110 ms in men or < 100 ms in women or;
  * Bradycardia with left bundle branch block and QRS duration > 140 ms in men or > 130 ms in women or;
  * Bradycardia with right bundle branch block and QRS duration > 130 ms in men or > 120 ms in women or;
  * Heart failure with left bundle branch block and QRS duration > 140 ms in men or >130 ms in women.
* Understands the nature of the study and is willing to comply with all study requirements.
* Provides written informed consent.
* A negative pregnancy test prior to the procedure for participants of child-bearing potential.

Exclusion Criteria:

* Complete AV block (3rd-degree AV block) without a stable escape rhythm or other circumstances where there is no measurable QRS.
* Subjects with a previous or current pacemaker or defibrillator implant.
* Anatomical or other conditions that may make a 12-lead ECG difficult to obtain, such as an allergy to components of the ECG pads, burns, open wounds, etc.
* Currently enrolled in another investigational device or drug trial that has not completed the active treatment phase and/or would conflict with this study.
* Other co-morbid condition(s) that could limit the participant's ability to participate in the study or to comply with study requirements or impact the scientific integrity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Different QRS duration requirements for male and female.
Study Population: Participants who are eligible for this study must have bradycardia or heart failure and are scheduled for pacemaker device implantation. Baseline ECG requirements must be met.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Predictive agreement between UHF-ECG and standard ECG | Pre-procedure
  Positive and negative predictive agreement between standard 12-lead ECG and UHF-ECG in discrimination of ventricular synchrony versus dyssynchrony with one recording per participant taken pre-procedure as evaluated by the core laboratory.

SECONDARY OUTCOMES:
Predictive agreement in dyssynchrony between UHF-ECG and standard ECG | Pre-procedure
  Predictive agreement of ventricular dyssynchrony and sidedness on the pre-procedure 12-lead ECG compared of UHF-ECG in participants with identified ventricular dyssynchrony.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - Peak Heart and Vascular, Avondale, Arizona
  - Banner Medical Center, Mesa, Arizona
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- St. Anne's University Hospital, Brno, Czechia
- Catherina Ziekenhuis, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plesinger F, Jurak P, Halamek J, Nejedly P, Leinveber P, Viscor I, Vondra V, McNitt S, Polonsky B, Moss AJ, Zareba W, Couderc JP. Ventricular Electrical Delay Measured From Body Surface ECGs Is Associated With Cardiac Resynchronization Therapy Response in Left Bundle Branch Block Patients From the MADIT-CRT Trial (Multicenter Automatic Defibrillator Implantation-Cardiac Resynchronization Therapy). Circ Arrhythm Electrophysiol. 2018 May;11(5):e005719. doi: 10.1161/CIRCEP.117.005719. Epub 2018 Apr 26. PMID 29700054
- [Background] Jurak P, Bear LR, Nguyen UC, Viscor I, Andrla P, Plesinger F, Halamek J, Vondra V, Abell E, Cluitmans MJM, Dubois R, Curila K, Leinveber P, Prinzen FW. 3-Dimensional ventricular electrical activation pattern assessed from a novel high-frequency electrocardiographic imaging technique: principles and clinical importance. Sci Rep. 2021 Jun 1;11(1):11469. doi: 10.1038/s41598-021-90963-4. PMID 34075135
- See also: sponsor website — http://www.vdimaging.com